## Official Title of the study:

Effect of Interventions Based on Acceptance and Commitment Therapy Administered to Parents of Special Needs Children on Their Levels of Psychological Resilience, Depression, Anxiety, Stress and Caregiver Burden: A randomised controlled trial

ClinicalTrials.gov Identifier: NCT04307706

**Date of the document:** 01.04.2019

## **ACT-based Intervention Study Protocol**

| Sessions | Aim | Time | Material | Interventions | Evaluations |
|---|---|---|---|---|---|
| Preparatory<br>Session | <ul> <li>Meeting and establishing therapeutic relationship</li> <li>Getting informed consent</li> <li>Explanation of the purpose of the training</li> <li>Collection of pre-test data</li> <li>Taking the participant's story</li> <li>Formulation through behavioral analysis</li> </ul> | 60 minutes | -A4 paper -Data collection tools (AAQ-II, RSA-21, DASS-21) -The Bull's Eye worksheet | <ul> <li>Applying Two Mountain metaphors</li> <li>Case formulation: Identifying excesses and shortcomings</li> </ul> | <ul> <li>Assessing whether the purpose of the training is understood</li> <li>Ending the session with feedback</li> </ul> |
| I. Session<br>Values: Clarifying<br>values | <ul> <li>Determining the interventions goals with the client</li> <li>Increasing awareness of her/his values, clarifying values, evaluations and trying to connect with her/his values.</li> </ul> | 60 minutes | -A small clipboard<br>-A4 paper<br>-Colorful pencils<br>-The Bull's Eye worksheet<br>-Values list / Value cards | <ul> <li>Clarifying values</li> <li>Apply the magic wand metaphor</li> <li>Breathing and mindfulness exercises</li> </ul> | ➤ Homework assignment: - Noticing what you are doing in line with your values - Breathing and mindfulness exercises ➤ Ending the session with feedback |
| II. Session Values and Creative hopelessness | <ul> <li>Setting the agenda by checking homework and summarizing the previous session</li> <li>Determining emotional control strategies</li> <li>To increase awareness of emotional control agenda</li> <li>Revealing dysfunctional behavior</li> </ul> | 60 minutes | -Rope or belt -A small clipboard -A4 paper | Forming of tried-and- tested solutions and their long-term effects. - Creative hopelessness intervention > Tug of war with a monster metaphor > Struggling in quicksand metaphor | ➤ Homework assignment: - Filling the tried-and-tested solutions and their long-term effects table - Keep a diary (until next session) ➤ Ending the session with feedback |
| III. Session Defusion | <ul> <li>Setting the agenda by checking homework and summarizing the previous session</li> <li>To see the real / real nature of the thoughts</li> <li>To react by considering the functionality of the thoughts, not their dictionary meanings</li> </ul> | 60 minutes | Notebook | <ul> <li>The leaves on a stream</li> <li>A master storyteller</li> <li>Letting it be:<br/>Singing and silly voices</li> </ul> | ➤ Homework assignment: - Practice the leaves on a stream exercise - Repeating the thought as singing and silly voices ➤ Ending the session with feedback |

| IV. Session Acceptance and Contact with the Present Moment | <ul> <li>Setting the agenda by checking homework and summarizing the previous session</li> <li>Allowing to experience painful personal experiences that serve their values</li> <li>To increase conscious awareness of the client's momentary experiences, to fully understand what is happening by bringing together important information about changing or maintaining behavior.</li> </ul> | 60<br>minutes | Notebook | AAAAAA | The struggle switch Demons on the Boat Mindful walking Time machine Breathing exercise Awareness five things | ➤ Homework assignment: - Recognizing when they struggle with their feelings and open up to them - Doing a work as 'mindful' - Mindful-breathing exercise for 10 minutes ➤ Ending the session with feedback |
|---|---|---|---|---|---|---|
| V. Session Self-as-context, Values and Committed Action: Doing what matters | <ul> <li>Setting the agenda by checking homework and summarizing the previous session</li> <li>Making a connection with the sense of self, independent of the client's thoughts and feelings, providing a safe and stable point of view for observing and accepting them.</li> <li>Transforming values into ongoing and progressive forms of action</li> </ul> | 60 minutes | Notebook | A A AA | The sky and the weather metaphor The Chessboard Metaphor Talking and listening Values and table of values commited action (to be created with parents) | ➤ Homework assignment: - Self-observation during mindful-practice - Take a step action on values - Noting what they did for their values in the created table ➤ Ending the session with feedback |
| VI. Session Values and Committed Action: Doing what matters | <ul> <li>Setting the agenda by checking homework and summarizing the previous session</li> <li>Transforming values into ongoing and progressive forms of action</li> <li>Enabling clients to reconnect with values the moment they move away from their values or lose the relationship</li> </ul> | 60 minutes | Notebook | A | Values and table of values commited action (to be created with parents) | ➤ Homework assignment: - Continuing with committed oriented actions as determined - Collection of post-test data - Informing for follow-up testing ➤ Ending the session with feedback |